CLINICAL TRIAL: NCT05707988
Title: Development and Evaluation of a Surgical Planning Tool for Urolithiasis Surgery: Kidney Stone Calculator
Brief Title: Kidney Stone Calculator
Acronym: KSC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP221171
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Urolithiasis
Keywords: Laser; Urolithiasis; Endoscopy; Ureteroscopy
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Urolithiasis is a frequent pathology, for which flexible ureteroscopy with endocorporeal laser lithotripsy has become the most frequently used surgical treatment. This procedure is limited to 90 minutes and will depend mainly on the total lithiasis volume. Knowing the duration of lithotripsy before the operation would allow to foresee situations of iterative procedures and to improve the patient's path (ambulatory or conventional surgery, work stoppage, optimization of operating times and operating room occupation times). "Kidney Stone Calculator" is a free tool capable of providing a calculi volumetry and predicting the duration of endocorporeal laser lithotripsy.

The main objective of this study would be to evaluate the performance of the Kidney Stone Calculator in estimating the duration of laser lithotripsy during flexible ureteroscopy for renal calculi, by analyzing the agreement between the estimated and actual lithotripsy durations, evaluated by an intraclass correlation coefficient and its 95% confidence interval Eligible patients will be those scheduled for flexible ureteroscopy for renal calculi described on a non-injected abdominopelvic scan. A total of 240 patients over a 15-month inclusion period is planned, with a follow-up time of 3 months.

DETAILED DESCRIPTION:
Urolithiasis is a common disease (10% of the general population). A quarter of patients will require surgery to treat a kidney stone. Ureteroscopy with endocorporeal laser lithotripsy is spreading and represents now the procedure of choice to treat a kidney stone. Its duration is variable and limited to 90min for infectious reasons. Having a tool to predict the duration of the procedure would allow to plan the patient's stay in the best possible way with a triple interest (patient, practitioner and administration).

"KIDNEY STONE CALCULATOR"(KSC) was developed to improve operative planning for lithiasis surgery. KSC estimates the total lithiasis volume from the patient's preoperative CT scan, using computer density segmentation, and then provides an estimate of the LLE duration (DEs) based on the computational density and laser parameters (energy, frequency, laser fiber diameter, laser type). Our KSC tool also allows the selection of laser parameters to optimize the duration of the computation fragmentation. These parameters could therefore also have an influence on the lithotripsy duration.

A first evaluation of KSC was performed in 2020 using operative data from 26 patients showing a small difference between the actual (Def) and estimated (Des) lithotripsy durations (median difference:14% (Q1-Q3(5.4-24.8);p = 0.36). The agreement between estimated and actual duration assessed by a CCI was 0.92 [0.78 - 0.97]. The duration of lithotripsy corresponded, together with the recovery time of the residual fragments, to half of the total operative time. Therefore, we would be able to predict the operative time with this tool. To date, this is the only study to estimate the duration of lithotripsy during an endoscopic kidney stone procedure.

We hypothesize a good concordance between estimated (Des) via KSC and actual (Def) lithotripsy durations during URS for renal calculi. This study will allow us to confirm the results of our pilot study and also to study the factors (patient (anatomy, number of stones and their positions and/or volumes, intraoperative), material used, experience of the operator) influencing Des.

Our study protocol plan to enroll 223 patients on 4 centers, on a prospective observational design.

This multicenter project in the Assistance Publique-Hôpitaux de Paris will be based on four Urology centers with a local manager:

* Tenon Hospital (Dr PANTHIER, Pr TRAXER)
* La Pitié-Salpétrière Hospital (Dr PINAR)
* Georges Pompidou European Hospital (Dr POINARD)
* Cochin Hospital (Dr ANRACT)

The Tenon team will be responsible for the local inclusions and for the coordination and support of the inclusions in the other centers. The principal investigators at La Pitié-Salpétrière, Hôpital Européen Georges Pompidou and Cochin will be responsible for the recruitment and inclusion of patients and for the postoperative follow-up according to the usual management in their center.

The estimated duration of each lithotripsy (Des) and of any residual stones after surgery will be determined centrally by Dr. Panthier, on the preoperative scans and on the scan performed for the postoperative follow-up consultation.

The local managers will be involved in the communication and valorization of this project in the form of a publication.

Patient recruitment procedures The overall management of the included patients will be in accordance with the usual management and recommendations.

Patients will be identified and recruited via the preoperative urology consultation of each center. Eligible patients will be informed of the study by the local investigator in charge of the patient, and the patient's non-objection will be collected during this consultation (or on the morning of the scheduled procedure if the patient wishes to have time to reflect).

The preoperative CT scan will be given to the surgeon and transmitted to the principal investigator to allow the latter to estimate the volume of lithiasis before the operation and to program the operation within 2 months following the preoperative consultation. The surgeon will have to record the laser parameters he intends to use (Energy (J), Frequency (Hz)) before the surgical procedure.

This observational study will not alter the usual management of patients, either preoperatively, intraoperatively or postoperatively. It consists of the collection of operative data, recorded in the operative report of a flexible ureteroscopy with endocorporeal laser lithotripsy (ELL), pre- and postoperative demographic and imaging data.

Patient follow-up schedule Procedure The patient will be operated by flexible ureteroscopy with endocorporeal laser lithotripsy within 2 months following the preoperative consultation.

The parameters of the procedure (duration, laser parameters and possible complications) will be recorded on a dedicated sheet provided for this purpose

Post-operative consultation The follow-up will be in accordance with the international recommendations with a consultation and a postoperative scan performed within 30 days following the procedure.

After the operation, the patients will be reviewed in a postoperative consultation (max. 30 days) for removal of the JJ probe.

The postoperative CT scan will determine :

* the absence of a residual fragment or
* reprogramming of a new operation (if residual fragments). The presence of residual fragments on the postoperative CT scan (bone window) is defined by the description of stones of 3mm or more in major axis.

Calculation of the Des

Before the procedure, the principal investigator will perform a volumetric evaluation of the stone by segmentation from the non-injected abdominopelvic CT scan in the bone window and an estimation of the lithotripsy duration according to the parameters chosen by the surgeon preoperatively on Kidney Stone Calculator. The same procedure will be performed with the intraoperative laser parameters chosen by the surgeon if they were different.

The estimation of the lithotripsy(Des) duration will be done before the operation and blinded to the surgeon.

In case of residual fragments on the postoperative CT scan, the volume of these stones will be subtracted from the preoperative lithiasis volume to adequately judge the effective duration of lithotripsy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* One or more kidney stones documented on a preoperative non-injected abdominopelvic CT scan
* scheduled for flexible ureteroscopy with endocorporeal laser lithotripsy
* using a reference laser (Holmium:YAG or Thulium Fiber)
* no opposition to the reuse of care data for research

Exclusion Criteria:

* Ureteral calculi
* Encrusted JJ stent
* Percutaneous surgical stone management
* Planned monobloc extraction of the stone
* Suspicion of struvite type stone (phosphasto-amoniacal-magnesium)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be defined as the population respecting the following criterias :
  Patient will be enrolled at the preoperative urologic consultation.
  Inclusion Criteria :
  * Age ≥ 18 years
  * One or more kidney stones documented on a preoperative non-injected abdominopelvic CT scan
  * scheduled for flexible ureteroscopy with endocorporeal laser lithotripsy
  * using a reference laser (Holmium:YAG or Thulium Fiber)
  * no opposition to the reuse of care data for research
  Exclusion Criteria :
  * Ureteral calculi
  * Encrusted JJ stent
  * Percutaneous surgical stone management
  * Planned monobloc extraction of the stone
  * Suspicion of struvite type stone (phosphasto-amoniacal-magnesium)
Sampling Method: Non-Probability Sample
Enrollment: 223 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Concordance | 3 months
  Concordance between estimated and actual laser lithotripsy times during flexible ureteroscopy for kidney stones, assessed by an intraclass correlation coefficient and its 95% confidence interval

SECONDARY OUTCOMES:
Correlation between Des and Def according to demographic, anatomical, number and types of calculi and their position, material | 3 months
  Suspected stone types will be defined based on their maximum density on the preoperative abdominopelvic CT and classified as follows:
  * Hard (density > 1000UH): Calcium oxalate monohydrate and phosphocalcic
  * Soft (density < 1000 HU): Uric acid/Calcium oxalate dihydrate/Cystine
Comparison of the surgeon's planned laser parameters and those used during the procedure for lithiasis fragmentation | 3 months
  comparison between the surgical notification absence of residual fragments at the end of lithotripsy (defined by a maximum diameter < 3mm according to current recommendations) with the assessment performed on the postoperative abdominopelvic CT scan.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric PANTHIER, MD, MSc, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Urology Department, Tenon Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided